CLINICAL TRIAL: NCT00299988
Title: A Placebo-controlled, Randomized, Double-Blind Phase II Clinical Study of Gammagard Intravenous Immunoglobulin (IVIg) for Treatment of Mild to Moderate Alzheimer's Disease
Brief Title: Phase II Study of Intravenous Immunoglobulin (IVIg) for Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Baxter BioScience (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 0512008265
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Results first posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-11

CONDITIONS: Alzheimer's Disease
Keywords: Immunotherapy; Amyloid beta protein; Antibodies; Alzheimer's; Dementia
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid; Dementia | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVIG (Experimental): ivig
  Interventions: Drug: Intravenous Immunoglobulin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Intravenous Immunoglobulin
  Arms: IVIG
Other: Placebo
  Arms: Placebo

SUMMARY:
The overall goal of this double-blind Phase II study is to evaluate the safety, efficacy and biological mechanisms of action of Intravenous Immunoglobulin (IVIg) in the treatment of mild to moderate stage Alzheimer's disease (AD). IVIg contains antibodies against the amyloid beta protein that is the central component of the AD senile plaque. It is hypothesized that IVIg treatment will reduce the levels of beta amyloid in the brain and improve cognitive abilities relative to placebo. A total of 24 patients with mild to moderate AD capable of giving informed consent will be randomly assigned to receive either IVIg (16 patients)or saline placebo (8 patients) for six months. This study includes comparison of four dosing regimens of IVIg. Cognitive, behavioral and functional measures will be collected at baseline, three months and six months of treatment. Plasma samples will be collected before and after infusions. Subjects will undergo a lumbar puncture before and after the six months of treatment for cerebrospinal fluid (CSF) biomarker analyses. In addition, Positron Emission Tomography (PET) imaging substudies will be performed at two time points during the study. Following the initial 6 month placebo-controlled period, all participants have the opportunity to receive IVIg for an additional 12 month period in an extension study.

DETAILED DESCRIPTION:
Abnormal processing of the beta-amyloid protein is thought to be an early and causative event in the pathogenesis of Alzheimer's disease (AD). Immunotherapy targeting beta amyloid (Aβ) has demonstrated a remarkable capacity to arrest and even reverse elements of AD brain pathology. Intravenous Immunoglobulin (IVIg) is a medication obtained from the pooled plasma of healthy human blood donors that contains natural anti-amyloid antibodies and exhibits potent central nervous system anti-inflammatory properties. IVIg has been FDA-approved and used for more than 25 years in patients with a variety of immune deficiency and autoimmune diseases and has an established safety record, but is not FDA-approved for the treatment of AD.

A total of 24 patients, males and females 50 years of age and older, with mild to moderate Alzheimer's disease (AD) will be enrolled in this research study. To be eligible, patients must meet the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria for probable AD. After written informed consent is obtained, subjects will go through a screening process to determine if he or she meets the inclusion criteria. Screening procedures include medical history, blood and urine tests, neurologic exam, chest x-ray and MRI. Women who want to take part in this study must either be post-menopausal, surgically sterilized or agree to avoid becoming pregnant during the entire period of their participation in this study.

To be eligible for this research study, patients must be taking a stable dose of an approved AD medication for at least 3 months prior to entering this study or be unable to take these medications. The design of this protocol is that of an add-on study and we will recommend patients continue to take any FDA-approved AD medications they are taking at study entry.

Subjects' participation in the study will last approximately 19 months, including screening and baseline procedures, treatment with study drug and a follow-up visit 1 ½ months after finishing treatment, plus a visit for blood tests 6 months after the last infusion in the study. This research study requires that the patient have another person, (such as a spouse, child, other relative, close friend, aide or other professional caregiver), who will accompany the patient to each clinic visit.

Subjects will be randomized to a treatment group for 6 months of infusions of IVIg or placebo. The treatment groups compare different doses and frequencies of treatment. Patients will have a 33% chance of receiving placebo.

Blood will be obtained from subjects every two weeks and examined in our research laboratories to obtain more information about IVIg's biological effects. Cerebrospinal fluid will be obtained by lumbar puncture twice over the course of the study for the same purpose. Patients will be asked to allow a portion of a blood sample to be used for Apolipoprotein E (APOE) testing and banked for genetic research testing related to AD and aging, but do not have to participate in the testing or allow their blood sample to be stored in order to take part in the study.

Cognitive testing will be carried out at baseline and every three months over a period of 18 months. Results of cognitive testing will constitute the primary endpoint of this study. Positron Emission Tomography (PET) imaging substudies will be performed at two time points during the study. Safety laboratories and assessments will be carried out at regular intervals. Subjects will not be responsible for any research study-related costs but will be responsible for the costs of evaluations required to establish diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of probable Alzheimer's disease (AD) of mild to moderate severity (as determined by a Mini Mental State Examination (MMSE) score of 14 - 26 inclusive).
2. Ability to give informed consent, designate a decision-maker or have an already recognized decision-maker (such as a legal guardian or health care proxy).
3. Ability to comply with testing and infusion regimen.
4. An able caregiver willing to participate (such as a spouse, child, other relative, close friend, aide or other professional caregiver closely involved in helping the patient take care of himself/herself).
5. Venous access suitable for repeated infusion and phlebotomy.
6. On stable doses of approved AD medications for at least 3 months.
7. As applicable, on stable doses of psychoactive medications (e.g. antidepressants, antipsychotics) for at least 6 weeks.
8. Neuroimaging performed after symptom onset consistent with the patient's diagnosis.
9. Clinical laboratory values within normal limits or if abnormal, judged clinically insignificant by the Principal Investigator.
10. Women who want to take part in this study must either be post-menopausal, surgically sterilized or agree to avoid becoming pregnant during the entire period of their participation in this study.

Exclusion Criteria:

1. Non-Alzheimer dementia.
2. Active renal disease.
3. Abnormally high serum viscosity levels.
4. Immunoglobulin A (IgA) deficiency.
5. Untreated congestive heart failure, unstable angina or a history of recent myocardial infarction.
6. Unstable arrhythmia.
7. Untreated or poorly controlled hypercholesterolemia.
8. Untreated or poorly controlled hypertension.
9. Poorly controlled diabetes.
10. Thrombosis (central or peripheral) in the past year.
11. Modified Hachinski score > 5.
12. Active cancer diagnosis, except basal cell carcinoma.
13. Active autoimmune or neuroimmunologic disorder.
14. History of IVIg treatment in past 6 months.
15. Untreated major depression or other major psychiatric disorders.
16. Known coagulopathy or platelet counts < 100,000.
17. Positive serology for Hepatitis B or C, or HIV.
18. Active migraines or frequent headaches (3 or more times per week).
19. Taking immunosuppressive drugs.
20. Chronic (more than thrice weekly) use of non-steroidal anti-inflammatory drugs (NSAIDs), excluding aspirin 81 milligrams daily.
21. Received an investigational treatment for AD within 3 months of study entry.
22. A history of or current disorder or disease that in a physician co-investigator's judgment may impede the subject's participation in the study, pose immoderate risk to the patient or confound the results of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-02; Primary Completion 2009-01 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman R Relkin, M.D., Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- IVIG: ivig
  Intravenous Immunoglobulin
Period: Overall Study
Arm/Group | IVIG | Placebo
Started | 16 | 8
Completed | 16 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- IVIG: Intravenous Immunoglobulin
- Placebo: placebo
- Total: Total of all reporting groups
Arm/Group | IVIG | Placebo | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 8 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 7 | 4 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: ADAS-Cog
Description: The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) is a brief neuropsychological assessment used to assess the severity of cognitive symptoms of dementia. It is one of the most widely used cognitive scales in clinical trials and is considered to be the "gold standard" for assessing antidementia treatments. The ADAS-Cog range from 0 to 70, where higher scores indicate greater cognitive dysfunction.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | IVIG | Placebo
Number analyzed (Participants) | 16 | 8
units on a scale | NA [NA to NA] — After extensive review of the records the actual calculations of the data cannot be located. | NA [NA to NA] — After extensive review of the records the actual calculations of the data cannot be located.

2. Primary Outcome: CGIC
Description: The Clinical Global Impression of Change focuses on clinicians' observations of change in the patient's cognitive, functional, and behavioral performance since the beginning of a trial. It relies on both direct examination of the patient and interview of informants. Unlike a targeted symptom scale, it takes into account a subject's overall function in the cognitive, behavioral and functional activity domains. Scoring is based on an interview with the caregiver and examination of the patient by an independent evaluator, without consulting other information such as cognitive test results. The CGIC range from 1 to 7, where 1=very much improved since the initiation of treatment; 4=no change from baseline; 7=very much worse since the initiation of treatment.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | IVIG | Placebo
Number analyzed (Participants) | 16 | 8
units on a scale | NA [NA to NA] — After extensive review of the records the actual calculations of the data cannot be located. | NA [NA to NA] — After extensive review of the records the actual calculations of the data cannot be located.

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Placebo: Placebo (no treatment)
Arm/Group | IVIG | Placebo
All-Cause Mortality (participants affected / at risk) | 10/16 | 4/8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8
Other Adverse Events (participants affected / at risk) | 0/16 | 0/8

LIMITATIONS AND CAVEATS:
The study was terminated due to the results from another phase III study with IVIG: PMC5409846, NCT00818662

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes